CLINICAL TRIAL: NCT01723891
Title: Study To Compare Safety and Pharmacokinetic Properties of Surfolase Capsule and HT-002-01 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hyundai Pharmaceutical Co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HT-002-01
Record Dates: First submitted 2012-11-06; First posted 2012-11-08 (Estimated); Last update posted 2012-11-08 (Estimated); Status verified 2012-11

CONDITIONS: Healthy

ARMS (2):
- Surfolase capsule & HT-002-01 (Active Comparator)
  Interventions: Drug: Surfolase capsule; Drug: HT-002-01
- HT-002-01 & Surfolase capsule (Active Comparator)
  Interventions: Drug: Surfolase capsule; Drug: HT-002-01

INTERVENTIONS:
Drug: Surfolase capsule
Drug: HT-002-01

SUMMARY:
Study to compare safety and pharmacokinetic properties of surfolase capsule and HT-002-01 after oral administration for one day in healthy male volunteer.

ELIGIBILITY:
Inclusion Criteria:

1. healthy male subjects between the age of 20 and 55 years with body mass index between 18.5 and 25
2. Volunteers without apriority of chronic disease
3. Volunteers must be in good health as determined by the investigator based on a detailed medical history, full physical examination, electrocardiogram, laboratory tests and urinalysis
4. Volunteers who comply with the protocol, understand and sign an informed consent

Exclusion Criteria:

1. Sensitive response to acebrophylline and xanthine
2. Galactose intolerance, Lapp lactase deficiency and Glucose-Galactose Malabsorption
3. Known history of renal, hepatic, respiratory, neurologic, endocrine, cardiac vascular and hematopoietic disease, especially gallstone
4. Known history of gastrointestinal disease which affects the absorption of medicine.
5. Excluded by screening tests
6. Upper limit of AST, ALT>1.25 times Upper limit of total bilirubin>1.5 times
7. Estimated GFR<80mL/min/1.73m2)
8. systolic blood pressure < 90 or > 150, diastolic blood pressure <50 or >100
9. Known history of drug abuse
10. caffeine>5cups/day, alcohol>210g/week, 10 more cigarettes/day
11. Use of any prescription drug within 14days or over-the-counter (OTC) medication within 7 days prior to dosing
12. Participation in any clinical investigation within 60 days prior to study start
13. Donation of blood within 60 days, donation of component blood within 30days
14. Judged by the investigators to be undesirable as subjects

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-11

PRIMARY OUTCOMES:
AUCt, Cmax

SECONDARY OUTCOMES:
AUCinf, Tmax, t1/2

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, Seoul, South Korea